CLINICAL TRIAL: NCT01255878
Title: The Efficacy of Gabapentine and Splint Therapy in Bruxers: a Randomized Clinical Trial
Brief Title: Comparative Evaluation of Gabapentine and Occlusal Splint in the Management of Sleep Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 87284
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Sleep Bruxism
Keywords: Sleep bruxism; Gabapentine; Occlusal splint; Polysomnography
MeSH Terms: conditions — Sleep Bruxism | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- stabilization splint (Experimental)
  Interventions: Device: occlusal stabilization splint
- Gabapentine (Experimental)
  Interventions: Drug: Gabapentine

INTERVENTIONS:
Device: occlusal stabilization splint
  Arms: stabilization splint
Drug: Gabapentine — 100 mg(1 capsule)three times per day for two months
  Arms: Gabapentine

SUMMARY:
Sleep bruxism (SB) is defined as a "stereotyped movement disorder characterized by grinding or clenching of the teeth during sleep" usually associated with sleep arousal. It might lead to abrasive tooth wear, hypermobility of teeth, tooth hypersensitivity, hypertrophy of the masticatory muscles and pain in the masticatory muscles.

Diagnostic procedures include clinical evaluation, ambulatory monitoring sleep laboratory investigations and others. The clinical approach comprises the patient's history, orofacial examination, and tooth wear classification.

There is no specific treatment for bruxism. Management of SB comprises psychological, orodental and pharmacological strategies.Orodental therapies, including soft vinyl mouth guards or stabilization bite splints, probably function more like protectors of the orofacial structures rather than actually diminishing bruxism.Drug treatment of sleep bruxism is controversial since different treatment strategies have resulted in suppression or exacerbation of this condition.

Based on the current data, central primary efferents are the major drivers of bruxism. Therefore centrally acting agents such as antiepileptic drugs which also affect the sleep structure, might be effective on SB.

In a case report of bruxism, anxiety and tremor, the authors suggested that anti-convulsant Gabapentine may be a useful treatment for patients with antidepressant-induced bruxism. However in the absence of definitive evidence, the appropiate treatment of SB is still a matter of debate.

The objective of the present study was to compare the treatment efficacy of occlusal stabilization splint and Gabapentine on SB, using polysomnographically determined outcome measures for the quantification of sleep bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and polysomnographic criteria of sleep bruxism according to the international classification of sleep disorders

Exclusion Criteria:

* Loss of more than two teeth and having removable prosthesis
* Presence of a major malocclusion
* Using any medication with a known influence on sleep structure or sleep bruxism
* Being diagnosed with psychological or neurotic disorders.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Azamsadat Madani, Dr, Study Director — Mashhad University of Medical Sciences; Nadia Hasanzadeh, Dr, Principal Investigator — Mashhad University of Medical Sciences; Hasan Azangoo, Dr, Principal Investigator — Mashhad University of Medical Sciences; Ebrahim Abdollahian, Dr, Study Director — Mashhad University of Medical Sciences
Locations (1):
- Mashhad University Of Medical Sciences, Mashhad, Khorasan Razavi, Iran

REFERENCES:
- [Background] Brown ES, Hong SC. Antidepressant-induced bruxism successfully treated with gabapentin. J Am Dent Assoc. 1999 Oct;130(10):1467-9. doi: 10.14219/jada.archive.1999.0057. PMID 10570590
- [Background] Dube C, Rompre PH, Manzini C, Guitard F, de Grandmont P, Lavigne GJ. Quantitative polygraphic controlled study on efficacy and safety of oral splint devices in tooth-grinding subjects. J Dent Res. 2004 May;83(5):398-403. doi: 10.1177/154405910408300509. PMID 15111632
- [Background] Foldvary-Schaefer N, De Leon Sanchez I, Karafa M, Mascha E, Dinner D, Morris HH. Gabapentin increases slow-wave sleep in normal adults. Epilepsia. 2002 Dec;43(12):1493-7. doi: 10.1046/j.1528-1157.2002.21002.x. PMID 12460250
- [Background] Kast RE. Tiagabine may reduce bruxism and associated temporomandibular joint pain. Anesth Prog. 2005 Fall;52(3):102-4. doi: 10.2344/0003-3006(2005)52[102:TMRBAA]2.0.CO;2. PMID 16252740
- [Background] Kato T, Thie NM, Huynh N, Miyawaki S, Lavigne GJ. Topical review: sleep bruxism and the role of peripheral sensory influences. J Orofac Pain. 2003 Summer;17(3):191-213. PMID 14520766
- [Background] Lavigne GJ, Khoury S, Abe S, Yamaguchi T, Raphael K. Bruxism physiology and pathology: an overview for clinicians. J Oral Rehabil. 2008 Jul;35(7):476-94. doi: 10.1111/j.1365-2842.2008.01881.x. PMID 18557915
- [Background] Lobbezoo F, Naeije M. Bruxism is mainly regulated centrally, not peripherally. J Oral Rehabil. 2001 Dec;28(12):1085-91. doi: 10.1046/j.1365-2842.2001.00839.x. PMID 11874505
- [Background] Placidi F, Mattia D, Romigi A, Bassetti MA, Spanedda F, Marciani MG. Gabapentin-induced modulation of interictal epileptiform activity related to different vigilance levels. Clin Neurophysiol. 2000 Sep;111(9):1637-42. doi: 10.1016/s1388-2457(00)00365-5. PMID 10964076
- [Background] Saletu A, Parapatics S, Anderer P, Matejka M, Saletu B. Controlled clinical, polysomnographic and psychometric studies on differences between sleep bruxers and controls and acute effects of clonazepam as compared with placebo. Eur Arch Psychiatry Clin Neurosci. 2010 Mar;260(2):163-74. doi: 10.1007/s00406-009-0034-0. Epub 2009 Jul 15. PMID 19603241
- [Background] Stapelmann H, Turp JC. The NTI-tss device for the therapy of bruxism, temporomandibular disorders, and headache - where do we stand? A qualitative systematic review of the literature. BMC Oral Health. 2008 Jul 29;8:22. doi: 10.1186/1472-6831-8-22. PMID 18662411
- [Background] Lavigne GJ, Rompre PH, Montplaisir JY. Sleep bruxism: validity of clinical research diagnostic criteria in a controlled polysomnographic study. J Dent Res. 1996 Jan;75(1):546-52. doi: 10.1177/00220345960750010601. PMID 8655758
- [Background] Lavigne GJ, Rompre PH, Poirier G, Huard H, Kato T, Montplaisir JY. Rhythmic masticatory muscle activity during sleep in humans. J Dent Res. 2001 Feb;80(2):443-8. doi: 10.1177/00220345010800020801. PMID 11332529